CLINICAL TRIAL: NCT00466557
Title: Genetic Association Mapping of Malaria Resistance in Anopheles Gambiae
Brief Title: Plasmodium Resistance in A. Gambiae
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 06-0084
Record Dates: First submitted 2007-04-26; First posted 2007-04-27 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2012-05

CONDITIONS: Malaria; Plasmodium Falciparum Malaria
Keywords: Malaria, Plasmodium falciparum, mosquito, Africa, Anopheles
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to find new ways to control malaria by looking at mosquitoes infected with the disease. Knowledge of the genetics that affect the spread of malaria by mosquitoes will help in developing control strategies. A small amount of blood from infected humans will be used to infect the mosquitoes. No contact will occur between the human subject and the mosquito. Study participants will be divided into 2 groups of 20, for a total of 40 children, ages 5-10, in Burkina Faso, West Africa. Each subject will be screened by finger-prick once per month, from June through October, until they reach a maximum age of 10. Two positive subjects of the 40 screened will be asked to donate about 1 teaspoon of blood, which will be used to feed and infect the mosquitoes. Study participants will be involved in study related procedures for a maximum of 5 years.

DETAILED DESCRIPTION:
Malaria is a blood-borne human disease, and is transmitted to mosquitoes in the bloodmeal, an obligatory step in human malaria transmission. This is a study of malaria parasites in the major mosquito vector of human malaria in Africa, Anopheles gambiae. The intent of the study is to develop modern forms of vector control that would specifically decrease disease transmission by targeting the vector. Genetic linkage mapping of the mosquito vector (Anopheles gambiae) in Africa has identified a small genomic region in the mosquito that controls most of the natural genetic variation for resistance to mosquito infection with the human malaria parasite (Plasmodium falciparum). In order to study the influence of mosquito vector genetics on transmission of malaria parasites, mosquitoes are exposed to malaria parasites and then the efficiency of parasite development within the mosquito is measured. The goal of the study is to promote and expand this non-transmitting subset of the vector population in order to decrease or interrupt human malaria transmission. The study focuses on the mosquito vector, not the human subjects infected with malaria. The reason for the use of human subjects is that 5cc of blood from human subjects naturally infected with malaria will be used to infect the mosquitoes by an indirect feeding method that involves a membrane feeding device. There will be no contact of human subjects with the mosquitoes. The blood-fed mosquitoes are the primary focus of this study, not human subjects. DNA extracted from mosquitoes that fed on the blood of human study subjects will be analyzed genetically by microsatellites and single-nucleotide polymorphisms (SNPs) to identify mosquito genes that control mosquito resistance to malaria parasites. The genetic analysis is of mosquito DNA, not DNA of the human subjects. At the time mosquitoes are analyzed, one week after the bloodmeal, there is no residual genetic, DNA, cellular, or any material of the human subject remaining within the mosquito, and thus no genetic or other information can derive from the human source, even accidentally. A secondary objective will be to identify naturally-occurring mechanisms of mosquito resistance to malaria infection in Burkina Faso. Mosquitoes that are not infected by malaria parasites do not transmit malaria. Research that identifies these genes for resistance may lead to a method for blocking the transmission of malaria. A total enrollment of 40 healthy volunteers, 5-10 years old, is planned at one site in Burkina Faso, West Africa. Malaria transmission occurs during the rainy season (June through October). There will be 2 experimental cycles per month from June through October (10 cycles per year). There will be two such groups of 20, for a total study size of 40. Each group of 20 will be screened for malaria in an alternating pattern, so each group of 20 is screened no more frequently than once per month during the malaria transmission season, for a total study duration of 5 years. One human subject with mature malaria gametocytes (the transmission stage infective to mosquitoes) will be identified the day before the projected experimental infection of mosquitoes. Blood (5 cc) will be drawn from the subject, which will occur no more frequently than once per month. Twenty subjects are screened for malaria parasites (by standard diagnosis) to insure finding at least one positive donor per cycle. The 5cc of blood is used to feed and infect mosquitoes, which are the subject of this study. Subject participation is approximately 5 months per year, for the total study duration of 5 years. A target sample size of 200 mosquitoes with a set of 150 markers will be analyzed in this study. A successful outcome of this study is genetic identification of mosquito genes controlling resistance and susceptibility to P. falciparum infection of the mosquitoes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 5-10 years old
2. No major diagnosable health problems (compared to local population)
3. Willing to participate in the study
4. Identified as having a malaria infection by blood film examination

Exclusion Criteria:

1. Outside the inclusion age group
2. Specific major diagnosable health problems
3. Not willing to participate in the study

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40
Dates: Start 2007-06; Primary Completion 2012-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre National de Recherche et de Formation sur le Paludisme, West Africa, Burkina Faso